CLINICAL TRIAL: NCT05135000
Title: A Randomized, Participant- and Investigator-blinded, Placebo-controlled Study to Investigate Efficacy, Safety, and Tolerability of LTP001 in Participants With Pulmonary Arterial Hypertension
Brief Title: Study of Efficacy and Safety of LTP001 in Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLTP001A12201
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LTP001 (Experimental): Participants received LTP001, 6 mg, oral capsules, once daily in the morning for approximately 24 weeks
  Interventions: Drug: LTP001
- Placebo (Placebo Comparator): Participants received LTP001 placebo capsules matching LTP001 orally once daily in the morning for approximately 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LTP001 — LTP001, 6 mg, was administered orally once daily in the morning
  Arms: LTP001
Drug: Placebo — Placebo to LTP001 was administered once daily in the morning
  Arms: Placebo

SUMMARY:
The purpose of this study was to explore the efficacy and safety of LTP001 in participants with pulmonary arterial hypertension (PAH) to determine if LTP001 had an adequate clinical profile to warrant further clinical development in this indication.

DETAILED DESCRIPTION:
This study was a non-confirmatory, randomized, participant- and investigator-blinded, placebo controlled trial evaluating the efficacy and safety of LTP001 on top of standard of care in participants with PAH.

The study included a screening period of up to 8 weeks, followed by a 24-week treatment phase with daily dosing and visits scheduled approximately every 4 weeks. One follow-up visit, which also served as the end-of-study visit, was conducted approximately 30 days after the conclusion of the treatment phase. The total duration of the study, from the beginning of the screening period to the end-of-study visit, was approximately 37 weeks.

A total of 44 participants were planned to be randomized in a 3:1 ratio to receive either LTP001 6 mg or placebo.

ELIGIBILITY:
Inclusion Criteria:

* History of PAH belonging to one of the following subgroups of the Clinical Classification Group 1 (WHO):

  * participants with idiopathic pulmonary arterial hypertension (IPAH)
  * Hereditary pulmonary arterial hypertension
  * Congenital heart disease (surgically repaired at least 12 months prior to screening)
  * drug or toxin induced (for example, anorexigen, or methamphetamine use).
* Resting mean pulmonary arterial pressure (mPAP) > 25 mmHg; pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure < 15 mmHg, as determined by right heart catheterization within 20 days of randomization.
* Pulmonary Vascular Resistance > 6 Wood units (480 dynes s/cm-5), as determined by right heart catheterization within 20 days of randomization.
* WHO Functional Class II-III
* 6MWD must be between 150 and 550 m (inclusive). The qualifying test needs to be within 20 days of randomization. To meet the above criterion additional six minute walk test (6MWT) may be performed up to a maximum of 3 tests in total prior to dosing; the minimal time difference between two tests should be at least 4 h.

  * Standard of care therapy which is stable at least 6 weeks prior to RHC and qualifying 6MWT assessment within 20 days of randomization. Standard of care includes one or more of the following treatments:
  * prostacyclin analogues and receptor agonists (if I.V., dose adjustments must be within 20% of initial stable dose)
  * endothelin receptor antagonists (ERAs)
  * phosphodiesterase type 5 inhibitors (PDE5i)
  * soluble guanylate cyclase (sGC) stimulators

Exclusion Criteria:

* Participants with pulmonary hypertension (PH) in the Clinical Classification Groups 2-5 (WHO), and any PAH Group 1 subgroups not covered by Inclusion Criterion #4.
* Participants with a history of left sided heart disease, chronic left sided heart failure, congenital or acquired valvular disease compromising left ventricular function and/or pulmonary venous hypertension or symptomatic coronary disease (non-symptomatic, revascularized coronary artery disease would be acceptable).
* Participants with obstructive lung disease defined as: FEV1/FVC < 60% and FEV1 < 60% of predicted value after bronchodilator administration as well as participants with moderate or severe restrictive lung disease: Total Lung Capacity < 70% of predicted value. Testing must have occurred within 24months of screening. If historical testing is not available, then lung function testing must be conducted during the screening period.
* Acute or chronic impairment (other than dyspnea), which would limit the ability to comply with study requirements, including interference with physical activity and execution of study procedures such as 6MWT (e.g., angina pectoris, claudication, musculoskeletal disorder, multiple sclerosis, need for walking aids).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (2):
  - Pulmonary Associates PA, Mesa, Arizona
  - Medical Univ of South Carolina, Charleston, South Carolina
- Novartis Investigative Site, Caba, Buenos Aires, Argentina
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Amsterdam, Netherlands
- Poland (3):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Wroclaw
- Spain (3):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2578

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 56 participants were screened for the study. Out of these, 47 participants were randomized.
Period: Overall Study
Arm/Group | LTP001 | Placebo
Started | 35 | 12
Completed | 26 | 9
Not Completed | 9 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study Terminated by Sponsor | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LTP001 | Placebo | Total
Number analyzed (Participants) | 35 | 12 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.3 (13.03) | 45.3 (13.78) | 45.3 (13.07)
Age, Customized [Number; unit: Participants]
  18 - <65 | 32 | 11 | 43
  65 - <85 | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 10 | 39
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 32 | 11 | 43
  American Indian or Alaska | 2 | 0 | 2
  Asian | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Right Heard Catheterization Pulmonary Vascular Resistance (PVR) at Week 25
Description: PVR was defined as the resistance against blood flow from the pulmonary artery to the left atrium measured in dyn.s.cm-5
Time Frame: Baseline, Week 25
Population: The pharmacodynamic (PD) analysis set included all participants with available PD data and no protocol deviations with a relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: dynes.sec.cm^-5
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 24 | 8
dynes.sec.cm^-5 | -1.175 (254.0792) | -49.685 (181.3745)

2. Secondary Outcome: Change From Baseline in Six Minute Walk Distance (6MWD)
Description: 6MWD test measures the distance that a patient can walk on a flat, hard surface in a period of 6 minutes
Time Frame: Baseline, Weeks 13 and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 30 | 10
meters
  Week 13 n=30,10 | 3.2 (42.45) | 7.4 (29.34)
  Week 25 n=28,10: number analyzed (Participants) | 28 | 10
  Week 25 n=28,10 | 10.4 (44.36) | 21.0 (32.33)

3. Secondary Outcome: Change From Baseline in Right Atrium (RA) Pressures at Week 25
Description: The Right Heart Catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including RA pressures.
Time Frame: Baseline, Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 26 | 9
mmHg | -0.4 (4.40) | -0.6 (0.73)

4. Secondary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure at Week 25
Description: Right heart catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including pulmonary capillary wedge pressure (PCWP).
Time Frame: Baseline, Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 24 | 9
mmHg | 0.2 (3.66) | 0.9 (2.26)

5. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure at Week 25
Description: Right heart catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including pulmonary artery pressure.
Time Frame: Baseline, Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 26 | 9
mmHg | 0.4 (8.55) | -0.6 (5.61)

6. Secondary Outcome: Change From Baseline in Average Cardiac Output (CO) at Week 25
Description: Right heart catheterization (RHC) assessment was performed to assess several hemodynamic variables in pulmonary hypertension, including cardiac output (CO).
Time Frame: Baseline, Week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 26 | 8
liters per minute | 0.067 (1.0772) | 0.493 (0.9075)

7. Secondary Outcome: Change From Baseline in Fractional Area Change (FAC)
Description: Key right ventricular (RV) function endpoints such as RV fractional area change (RV FAC) were assessed with echocardiography.
Time Frame: Baseline, Weeks 5, 13, and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 31 | 10
percent
  Week 5 n=31,9: number analyzed (Participants) | 31 | 9
  Week 5 n=31,9 | 0.35 (6.944) | 0.92 (5.622)
  Week 13 n=29,10: number analyzed (Participants) | 29 | 10
  Week 13 n=29,10 | -1.19 (6.424) | 2.62 (4.417)
  Week 25 n=26,8: number analyzed (Participants) | 26 | 8
  Week 25 n=26,8 | -1.85 (5.412) | -1.45 (7.532)

8. Secondary Outcome: Change From Baseline in Peak Velocity of Excursion (RV S')
Description: Key right ventricular (RV) function per echocardiography. The terms Tricuspid Annular Systolic Velocity (TASV) and Peak Velocity of Excursion (RV S') are synonymous in echocardiography to describe the peak systolic velocity of the lateral tricuspid annulus. Including both TASV and RV S' as separate secondary endpoints was an oversight in the protocol as the data, calculation, and analyses for both (TASV and RV S') are identical. Therefore, the TASV and RV S' data in this results disclosure are the same.
Time Frame: Baseline, Weeks 5, 13, and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 33 | 11
centimeters per second
  Week 5 n=33,11 | 0.2 (2.14) | -0.4 (1.50)
  Week 13 n=32,11: number analyzed (Participants) | 32 | 11
  Week 13 n=32,11 | -0.2 (2.38) | -0.5 (1.63)
  Week 25 n=26,9: number analyzed (Participants) | 26 | 9
  Week 25 n=26,9 | 0.4 (2.28) | -1.0 (3.00)

9. Secondary Outcome: Change From Baseline in Tricuspid Annular Plane Systolic Excursion (TAPSE)
Description: Key right ventricular (RV) function endpoints such as tricuspid annular plane systolic excursion (TAPSE) were assessed with echocardiography.
Time Frame: Baseline, Weeks 5, 13, and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 33 | 11
centimeters
  Week 5 n=33,11 | 0.061 (0.3181) | 0.042 (0.3383)
  Week 13 n=31,11: number analyzed (Participants) | 31 | 11
  Week 13 n=31,11 | -0.026 (0.2594) | 0.100 (0.2933)
  Week 25 n=27,9: number analyzed (Participants) | 27 | 9
  Week 25 n=27,9 | 0.015 (0.3697) | -0.067 (0.2121)

10. Secondary Outcome: Change From Baseline in Tricuspid Annular Systolic Velocity (TASV)
Description: Key right ventricular (RV) function endpoints such as tricuspid annular systolic velocity (TASV) were assessed with echocardiography.
Time Frame: Baseline, Weeks 5, 13 and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 33 | 11
centimeters per second
  Week 5 n=33,11 | 0.2 (2.14) | -0.4 (1.50)
  Week 13 n=32,11: number analyzed (Participants) | 32 | 11
  Week 13 n=32,11 | -0.2 (2.38) | -0.5 (1.63)
  Week 25 n=26,9: number analyzed (Participants) | 26 | 9
  Week 25 n=26,9 | 0.4 (2.28) | -1.0 (3.00)

11. Secondary Outcome: Change From Baseline in EmPHasis-10
Description: emPHasis-10 is a questionnaire with 10 questions designed to determine how pulmonary hypertension affects a participant's life. Each item is scored on a scale of 0 to 5, with a total score ranging from 0 to 50. A higher score indicates worse quality of life.
Time Frame: Baseline, Weeks 13 and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 21 | 9
score
  Week 13 n=21,9 | -1.490 (5.7108) | -3.622 (3.1712)
  Week 25 n=17,9: number analyzed (Participants) | 17 | 9
  Week 25 n=17,9 | -4.972 (8.7643) | -3.000 (4.2961)

12. Secondary Outcome: Change From Baseline in Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT)
Description: PAH-SYMPACT is a questionnaire used to assess pulmonary arterial hypertension symptoms and their impact. Individual item scores range from 0 to 4. Total score is calculated as the sum of the scores for the individual items divided by the number of items. A higher score indicates more severe symptoms/impacts.
Time Frame: Baseline, Weeks 13 and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 11 | 4
score
  Week 13 | -1.452 (6.3897) | -3.545 (3.2693)
  Week 25 | -0.680 (5.7304) | -4.220 (6.1990)

13. Secondary Outcome: Maximum Observed Blood Concentrations (Cmax) for LTP001
Description: The maximum (peak) observed blood drug concentration after single dose administration.
Time Frame: Day 1 and Week 25 at 15, 45, and 120 minutes post-dose
Population: The pharmacokinetic (PK) analysis set included all participants with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received any study drug, and without protocol deviations that impacted PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 30 | 0
ng/mL
  Day 1 | 38.6 (58.2) |
  Week 25: number analyzed (Participants) | 23 | 0
  Week 25 | 39.2 (54.7) |

14. Secondary Outcome: Time to Reach Maximum Blood Concentrations (Tmax) of LTP001
Description: The time to reach maximum (peak) blood drug concentration after single dose administration.
Time Frame: Day 1 and Week 25 at 15, 45, and 120 minutes post-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 30 | 0
hours
  Day 1 | 1.05 (56.6) |
  Week 25: number analyzed (Participants) | 23 | 0
  Week 25 | 0.979 (68.8) |

15. Secondary Outcome: Time to Clinical Worsening
Description: Time to any of the following:
  * Death
  * Hospital stay greater than 24 hours due to worsening of pulmonary arterial hypertension
  * Worsening of PAH resulting in need for lung transplantation or balloon atrial septostomy
  * Initiation of parenteral prostanoid therapy, initiation of oxygen therapy, initiation of any other pulmonary arterial hypertension-specific therapies or need for increase of diuretics for more than 4 weeks due to worsening of pulmonary arterial hypertension
  * Significant drop in six minute walk distance
Time Frame: Baseline up to approximately 30 weeks
Population: The pharmacodynamic (PD) analysis set included all participants with available PD data and no protocol deviations with a relevant impact on PD data. Participants without the event were considered as censored at the end of the time at risk.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 34 | 12
days | 211.0 [174.0 to NA] — The upper limit of 95% CI was not calculable due to an insufficient number of participants with events. | 175.0 [174.0 to NA] — The upper limit of 95% CI was not calculable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: LTP001 vs Placebo; Test type: Other; p = 0.6843, Log Rank; Cox Proportional Hazard = 0.7, 80% CI 2-sided [0.2 to 2.8]

16. Secondary Outcome: Change From Baseline in N-terminal Fragment of the Prohormone B-type Natriuretic Peptide (NT-ProBNP)
Description: NT-proBNP is a blood biomarker to assess right ventricular distress.
Time Frame: Baseline to Week 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picomoles per liter
Arm/Group | LTP001 | Placebo
Number analyzed (Participants) | 27 | 11
picomoles per liter | 4.609 (52.9047) | -7.918 (21.9731)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 241 days.
Groups:
- Total: Total
Arm/Group | LTP001 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/12 | 0/47
Serious Adverse Events (participants affected / at risk) | 5/35 | 2/12 | 7/47
Other Adverse Events (participants affected / at risk) | 20/35 | 7/12 | 27/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LTP001 (N=35) | Placebo (N=12) | Total (N=47)
Right ventricular failure (Cardiac disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LTP001 (N=35) | Placebo (N=12) | Total (N=47)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 3 | 1 | 4
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 1 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Asthenia (General disorders and administration site conditions) | 2 | 0 | 2
Chest discomfort (General disorders and administration site conditions) | 0 | 1 | 1
Fatigue (General disorders and administration site conditions) | 2 | 1 | 3
Influenza like illness (General disorders and administration site conditions) | 1 | 1 | 2
Peripheral swelling (General disorders and administration site conditions) | 2 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2
Respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 6 | 0 | 6
Presyncope (Nervous system disorders) | 2 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05135000/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT05135000/SAP_001.pdf